CLINICAL TRIAL: NCT05271539
Title: Comparative Study of the Efficacy of Intravitreal Ranibizumab Versus Its Combination With Commercial Dexamethasone in The Treatment of Diabetic Macular Edema
Brief Title: Intravitreal Ranibizumab Versus Its Combination With Dexamethasone in The Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, khaled gamal abueleinen, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-278-2020
Record Dates: First submitted 2022-02-15; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Intervention Model Description: The first group received 3 monthly intravitreal injections of 0.5 mg in 0.05 mL ranibizumab alone (Lucentis, by Novartis), aspirated from vial through 5-micron sterile filter needle (19-gauge × 1-1/2 inch), with a 1-mL syringe and injected through a 30-gauge × ½ inch sterile injection needle. While the second group received monthly intravitreal injections of the same dose of ranibizumab combined with 0.4 mg in 0.1 ml dexamethasone (Dexamethasone sodium phosphate, Amriya Pharmaceuticals, Cairo, Egypt) in a separate 1ml syringe with 27- gauge × ½ inch sterile injection needle, followed by 2 Intravitreal ranibizumab, 1 month apart (with dexamethasone if follow up OCT shows less than 10% improvement from baseline i.e., PRN).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The first group, Lucentis alone group (Active Comparator): The first group received 3 monthly intravitreal injections of 0.5 mg in 0.05 mL ranibizumab alone (Lucentis, by Novartis), aspirated from vial through 5-micron sterile filter needle (19-gauge × 1-1/2 inch), with a 1-mL syringe and injected through a 30-gauge × ½ inch sterile injection needle.
  Interventions: Drug: Lucentis alone group
- The second group, Lucentis dexamethasone group (Active Comparator): The second group received monthly intravitreal injections of the same dose of ranibizumab combined with 0.4 mg in 0.1 ml dexamethasone (Dexamethasone sodium phosphate, Amriya Pharmaceuticals, Cairo, Egypt) in a separate 1ml syringe with 27- gauge × ½ inch sterile injection needle, followed by 2 Intravitreal ranibizumab, 1 month apart (with dexamethasone if follow up OCT shows less than 10% improvement from baseline i.e., PRN).
  Interventions: Drug: Lucentis dexamethasone group

INTERVENTIONS:
Drug: Lucentis alone group — The Lucentis alone group received 3 monthly intravitreal injections of lucentis alone or less than 3 injections if the central foveal thickness reached 250 microns
  Arms: The first group, Lucentis alone group
Drug: Lucentis dexamethasone group — Lucentis dexamethasone group received intravitreal injections of combination of both lucentis and commercial dexamethasone. the second group received monthly intravitreal injections of the same dose of ranibizumab combined with 0.4 mg in 0.1 ml dexamethasone (Dexamethasone sodium phosphate, Amriya Pharmaceuticals, Cairo, Egypt) in a separate 1ml syringe with 27- gauge × ½ inch sterile injection needle, followed by 2 Intravitreal ranibizumab, 1 month apart (with dexamethasone if follow up OCT shows less than 10% improvement from baseline i.e., PRN). Treatment was stopped when CMT improved below 250 µ.
  Arms: The second group, Lucentis dexamethasone group

SUMMARY:
Intravitreal ranibizumab alone was Compared to adding dexamethasone to ranibizumab regarding central macular thickness, the visual acuity and the number of intravitreal injections needed to achieve the same effect on CMT and BCVA at the end of the 6 months duration of the study. Any significant change in final IOP, compared to baseline, in either group is reported.

DETAILED DESCRIPTION:
This prospective randomized study measures the changes in central macular thickness, best corrected visual acuity and IOP in diabetic macular edema before and after the intravitreal injection of ranibizumab and dexamethasone, compared to ranibizumab alone, the current gold standard of care for diabetic macular edema.

Study participants were randomized into 2 groups: the first group received 3 Intravitreal injections of ranibizumab alone 1 month apart. While the second group received 1 Intravitreal injection of a combination of ranibizumab and 0.4 mg in 0.1 ml dexamethasone followed by 2 Intravitreal ranibizumab, 1 month apart (with dexamethasone if follow up OCT shows less than 10% improvement from baseline). Treatment was stopped when the treated eye achieved a central macular thickness of 250 microns or less with no focal parafoveal edema.

Final recorded central macular thickness in both groups compared to the baseline. By the end of the follow up period.

Final visual acuity was assessed in both groups compared to the baseline Change in final IOP, compared to baseline, in ranibizumab group and ranibizumab with dexamethasone group.

. The number of injections needed to achieve the same effect on CMT and BCVA.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema with central macular thickness of 300 μm or greater (as measured by spectral domain optical coherence tomography [OCT]).
* Best corrected visual acuity of 6/12 or less.

Exclusion Criteria:

* ● History of any treatment for DME (including grid or focal laser photocoagulation) within the last 6 months

  * History of panretinal photocoagulation within the last 6 months.
  * PDR as indicated with Fluorescein Angiography as it will require PRP which may affect DME.
  * Macular ischemia, as indicated with Fluorescein Angiography.
  * Cataract surgery within three months or cataract that requires surgical intervention during the follow-up period.
  * Pseudophakia with Irvine Gass syndrome, as indicated with Fluorescein Angiography.
  * Vitreomacular traction syndrome.
  * Other causes of macular edema (eg. CRVO, CNV, uveitis, etc).
  * Glaucoma, whether suspected or confirmed.
  * Significant media opacity.
  * Patients with ocular or periocular infections, or infection in the other eye
  * Signs of Active or resolved uveitis and intraocular inflammation.
  * Bad diabetic control as indicated by HbA1C >8.
  * Renal impairment, hepatic impairment, or congestive heart failure.
  * History of cardiovascular insult or stroke.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Central foveal thickness | 6 months after the first injection
  Central foveal thickness in microns measured by OCT
BCVA (Decimal) | 6 months after the first injection
  Best corrected visual acuity measured on Snellen chart in Decimal form
The number of injections | over 6 months duration of the study
  The total number of injections in each Arm group

SECONDARY OUTCOMES:
IOP | 6 months after the first injection
  Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Khaled G Abueleinen, MD, PhD, Principal Investigator — Ophthalmology department, Faculty of Medicine Cairo University
Locations (1):
- Khaled G Abueleinen, Giza, Cairo Governorate, Egypt

REFERENCES:
- [Background] Maturi RK, Glassman AR, Liu D, Beck RW, Bhavsar AR, Bressler NM, Jampol LM, Melia M, Punjabi OS, Salehi-Had H, Sun JK; Diabetic Retinopathy Clinical Research Network. Effect of Adding Dexamethasone to Continued Ranibizumab Treatment in Patients With Persistent Diabetic Macular Edema: A DRCR Network Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jan 1;136(1):29-38. doi: 10.1001/jamaophthalmol.2017.4914. PMID 29127949